CLINICAL TRIAL: NCT05185089
Title: A Double-Blind, Randomised, Placebo Controlled, Two Period Cross-Over Study to Evaluate the Efficacy and Safety of Orvepitant in Chronic Cough in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Efficacy and Safety Study of Orvepitant for Chronic Cough in Patients With Idiopathic Pulmonary Fibrosis
Acronym: IPF-COMFORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nerre Therapeutics Ltd. (Industry)
Collaborators: Pharm-Olam International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORV-PF-01
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Cough; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Cough; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Orvepitant 30mg (Experimental): Orvepitant 30mg tablet once daily for 4 weeks
  Interventions: Drug: Orvepitant Maleate
- Orvepitant 10mg (Experimental): Orvepitant 10mg tablet once daily for 4 weeks
  Interventions: Drug: Orvepitant Maleate
- Placebo (Placebo Comparator): Placebo tablet once daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orvepitant Maleate — Orvepitant tablets 30mg or 10mg
  Arms: Orvepitant 10mg; Orvepitant 30mg
Drug: Placebo — Placebo tablets to match orvepitant 30mg and 10mg tablets
  Arms: Placebo

SUMMARY:
ORV-PF-01 is a two way, placebo controlled, cross-over study, to evaluate the effect of two doses of orvepitant on cough in patients with IPF.

DETAILED DESCRIPTION:
The study will be a multi-center, double-blind, randomised, placebo-controlled 2-period cross-over study in subjects with chronic cough due to idiopathic pulmonary fibrosis (IPF).

Subjects will participate in one of two cohorts (Cohort 1 and Cohort 2). Cohort 1 will evaluate a 30 mg orvepitant dose and Cohort 2 the 10 mg dose. Within each cohort, subjects will be randomised to receive either orvepitant or placebo in the first treatment period (Treatment Period A) followed by the alternate treatment in Treatment Period B. There will be a wash-out period of 3 weeks between the two treatment periods. Subjects will be randomised 1:1 to each of the two treatment orders and 1:1 to each cohort.

Subjects will enter a screening period of between 14 and 28 days to determine eligibility. Eligible subjects will be randomised at the Baseline visit and will participate in two identical 28 day treatment periods with the wash-out period between them. There will be a total of 8 visits including the Screening, Baseline and final Follow-up visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of IPF established according to the 2018 or 2022 joint ATS/ERS/JRS/ALAT Clinical Practice Guideline
* FEV1/FVC ratio ≥0.65 at the screening visit
* Haemoglobin-corrected diffusion capacity of carbon monoxide (Hb-corrected DLCO) ≥25% within 12 months of the screening visit
* Arterial oxygen saturation on room air or oxygen ≥90% at Screening
* Life expectancy of at least 12 months
* Cough that is attributed to IPF, which has not responded to anti-tussive treatment, and which has been present for at least 8 weeks prior to Screening
* Mean daily IPF Coughing Severity Scale score ≥5 (after rounding) during the second week of the baseline assessment period

Key Exclusion Criteria:

* Recent respiratory tract infection (<8 weeks prior to Screening)
* Recent acute exacerbation of IPF (<8 weeks prior to Screening)
* Current smokers or ex-smokers with <6 months' abstinence prior to Screening
* Emphysema ≥50% on high-resolution computed tomography, or the extent of emphysema is greater than the extent of fibrosis according to the reported results of the most recent scan
* Mean early morning cough scale score ≥5 and rest of the day cough scale score <5 (after rounding) during the second week of the baseline assessment period (assessed at Visit 2)
* Cough that is predominantly productive in nature and attributable to lung pathology such as chronic bronchitis or bronchiectasis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. S. Birring, MB ChB, MD, Principal Investigator — Department of Respiratory Medicine, King's College Hospital, London UK
Locations (37):
- United States (16):
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Loyola University Chicago, Maywood, Illinois
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - American Health Research, Charlotte, North Carolina
  - PulmonIx, LLC, Greensboro, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University, Dallas, Texas
  - Clear Lake Health, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
- Netherlands (4):
  - Zuyderland Medical Centre, Heerlen
  - Sint Antonius Hospital, Nieuwegein
  - Erasmus University Medical Centre, Rotterdam
  - Isala Ziekenhuis, Zwolle
- United Kingdom (17):
  - Royal Berkshire Hospital, Reading, Berkshire
  - Castle Hill Hospital, Cottingham, Hull
  - MAC Clinical Research, Prescot, Merseyside
  - Antrim Area Hospital, Antrim, Northern Ireland
  - Altnagelvin Area Hospital, Londonderry, Northern Ireland
  - Churchill Hospital, Headington, Oxford
  - Perth Royal Infirmary, Perth, Perth and Kinross
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - MAC Clinical Research, Barnsley, South Yorkshire
  - MAC Clinical Research, Leeds, West Yorkshire
  - Heartlands Hospital, Birmingham
  - Royal Papworth Hospital, Cambridge
  - Royal Devon and Exeter Hospital, Exeter
  - Guy's Hospital, London
  - MAC Clinical Research, Manchester
  - Nottingham City Hospital, Nottingham
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 participants were enrolled into the study. 40 were randomised to the orvepitant 10 mg cohort and 40 to the orvepitant 30 mg cohort.
Pre-assignment Details: This was a crossover study so each participant was to receive both orvepitant and placebo.
Groups:
- Placebo first, then orvepitant 10 mg: Participants first received placebo once-daily (one tablet each evening, matching orvepitant 10 mg) for 4 weeks (Period A). After a washout period of 3 weeks, they then received orvepitant 10mg once-daily (one tablet each evening) for 4 weeks (Period B).
- Orvepitant 10 mg first, then placebo: Participants first received orvepitant 10mg once-daily (one tablet each evening) for 4 weeks (Period A). After a washout period of 3 weeks, they then received placebo once-daily (one tablet each evening, matching orvepitant 10 mg) for 4 weeks (Period B).
- Placebo first, then orvepitant 30 mg: Participants first received placebo once-daily (one tablet each evening, matching orvepitant 30 mg) for 4 weeks (Period A). After a washout period of 3 weeks, they then received orvepitant 30mg once-daily (one tablet each evening) for 4 weeks (Period B).
- Orvepitant 30 mg first, then placebo: Participants first received orvepitant 30mg once-daily (one tablet each evening) for 4 weeks (Period A). After a washout period of 3 weeks, they then received placebo once-daily (one tablet each evening, matching orvepitant 30 mg) for 4 weeks (Period B).
Period: First Intervention (4 weeks)
Arm/Group | Placebo first, then orvepitant 10 mg | Orvepitant 10 mg first, then placebo | Placebo first, then orvepitant 30 mg | Orvepitant 30 mg first, then placebo
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 19
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout (3 weeks)
Arm/Group | Placebo first, then orvepitant 10 mg | Orvepitant 10 mg first, then placebo | Placebo first, then orvepitant 30 mg | Orvepitant 30 mg first, then placebo
Started | 20 | 20 | 20 | 19
Completed | 20 | 20 | 20 | 19
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (4 weeks)
Arm/Group | Placebo first, then orvepitant 10 mg | Orvepitant 10 mg first, then placebo | Placebo first, then orvepitant 30 mg | Orvepitant 30 mg first, then placebo
Started | 20 | 20 | 20 | 19
Completed | 19 | 19 (The SAE that resulted in death started during the washout period after receiving orvepitant 10 mg so fatal SAE reported in 'Orv 10 mg' arm. However, the participant died during the second intervention while receiving placebo so death reported in the 'Placebo (10 mg cohort)' arm.) | 20 | 19
Not Completed | 1 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a crossover study so participants were to receive both orvepitant and placebo.
Groups:
- Orvepitant 10 mg Cohort: Participants randomised to the orvepitant 10 mg cohort. They were randomised to receive either orvepitant 10 mg or placebo in the first treatment period (Treatment Period A), followed by the alternate treatment in Treatment Period B.
- Orvepitant 30 mg Cohort: Participants randomised to the orvepitant 30 mg cohort. They were randomised to receive either orvepitant 30 mg or placebo in the first treatment period (Treatment Period A), followed by the alternate treatment in Treatment Period B.
- Total: Total of all reporting groups
Arm/Group | Orvepitant 10 mg Cohort | Orvepitant 30 mg Cohort | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (6.55) | 72.4 (7.79) | 71.9 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 30 | 29 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 37 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 37 | 37 | 74
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Weekly Average of the Daily Idiopathic Pulmonary Fibrosis Coughing Severity Scale (IPF CSS)
Description: A numerical rating scale from 0 (no coughing) to 10 (coughing as bad as you can imagine) for coughing severity in the last 24 hours
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Placebo (10 mg Cohort): Placebo once-daily for 4 weeks in either Period A or Period B (subjects assigned to orvepitant 10mg cohort)
- Orvepitant 10 mg: Orvepitant 10 mg once-daily for 4 weeks in either Period A or Period B
- Placebo (30 mg Cohort): Placebo once-daily for 4 weeks in either Period A or Period B (subjects assigned to orvepitant 30mg cohort)
- Orvepitant 30 mg: Orvepitant 30 mg once-daily for 4 weeks in either Period A or Period B
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | -0.69 (1.583) | -0.66 (1.276) | -0.26 (1.155) | -0.85 (1.465)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.989, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.62 to 0.63], Standard Error of Mean 0.305
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.054, ANCOVA; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.16 to 0.01], Standard Error of Mean 0.293

2. Secondary Outcome: Mean Change From Baseline in Weekly Average of the Early Morning IPF Coughing Severity Scale
Description: A numerical rating scale from 0 (no coughing) to 10 (coughing as bad as you can imagine) for coughing severity first thing in the morning
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | -0.57 (1.505) | -0.51 (1.199) | -0.49 (1.184) | -1.08 (1.627)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.872, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.52 to 0.62], Standard Error of Mean 0.280
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.041, ANCOVA; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.14 to -0.02], Standard Error of Mean 0.276

3. Secondary Outcome: Mean Change From Baseline in Weekly Average of the Rest of the Day IPF Coughing Severity Scale
Description: A numerical rating scale from 0 (no coughing) to 10 (coughing as bad as you can imagine) for severity of any other coughing during the last 24 hours, excluding coughing first thing in the morning
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | -0.62 (1.477) | -0.62 (1.306) | -0.44 (1.117) | -0.80 (1.528)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.991, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.61 to 0.60], Standard Error of Mean 0.303
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.215, ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.97 to 0.22], Standard Error of Mean 0.298

4. Secondary Outcome: Mean Change From Baseline in Weekly Average of the Daily Urge to Cough Scale
Description: A numerical rating scale from 0 (no urge to cough) to 10 (urge to cough as bad as you can imagine) for severity of urge to cough in the last 24 hours
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | -0.46 (1.517) | -0.63 (1.209) | -0.30 (0.974) | -0.76 (1.400)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.639, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.73 to 0.45], Standard Error of Mean 0.291
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.092, ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.00 to 0.08], Standard Error of Mean 0.271

5. Secondary Outcome: Mean Change From Baseline in Weekly Average of the Daily Cough Frequency Scale
Description: A 5-point verbal rating scale for cough frequency over the last 24 hours with response options from 'never' to 'all the time'. The verbal responses were converted to a number (0 = never, 4 = all the time).
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | -0.20 (0.574) | -0.15 (0.543) | -0.06 (0.369) | -0.29 (0.462)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.650, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.17 to 0.26], Standard Error of Mean 0.104
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.41 to -0.06], Standard Error of Mean 0.085

6. Secondary Outcome: Mean Change From Baseline in Weekly Average of the Daily Dyspnoea Scale
Description: A numerical rating scale from 0 (no shortness of breath) to 10 (shortness of breath as bad as you can imagine) for severity of shortness of breath in the last 24 hours
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | -0.26 (1.192) | -0.22 (0.988) | 0.00 (0.764) | -0.44 (1.060)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.856, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.44 to 0.53], Standard Error of Mean 0.240
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.036, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.87 to -0.03], Standard Error of Mean 0.210

7. Secondary Outcome: Mean Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score
Description: The LCQ is a 19-item questionnaire that assesses cough-related Quality-of-Life. It has three domains (physical, psychological and social). The total score range is 3-21 and domain scores each range from 1-7; a higher score indicates a better Quality-of-Life. This outcome measure is the mean change from Baseline to Week 4 in the total score.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | 1.07 (2.218) | 1.27 (2.187) | 0.14 (2.724) | 1.60 (2.353)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.678, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.73 to 1.11], Standard Error of Mean 0.462
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.025, ANCOVA; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [0.16 to 2.31], Standard Error of Mean 0.525

8. Secondary Outcome: Mean Change From Baseline in Leicester Cough Questionnaire (LCQ) Physical Domain Score
Description: The LCQ is a 19-item questionnaire that assesses cough-related Quality-of-Life. It has three domains (physical, psychological and social). The total score range is 3-21 and domain scores each range from 1-7; a higher score indicates a better Quality-of-Life. This outcome measure is the mean change from Baseline to Week 4 in the physical domain score.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | 0.18 (0.656) | 0.26 (0.717) | 0.06 (0.750) | 0.36 (0.638)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.633, ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.22 to 0.35], Standard Error of Mean 0.143
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.063, ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.02 to 0.56], Standard Error of Mean 0.139

9. Secondary Outcome: Mean Change From Baseline in Leicester Cough Questionnaire (LCQ) Psychological Domain Score
Description: The LCQ is a 19-item questionnaire that assesses cough-related Quality-of-Life. It has three domains (physical, psychological and social). The total score range is 3-21 and domain scores each range from 1-7; a higher score indicates a better Quality-of-Life. This outcome measure is the mean change from Baseline to Week 4 in the psychological domain score.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | 0.57 (0.935) | 0.47 (0.906) | 0.12 (1.004) | 0.63 (0.984)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.732, ANCOVA; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.44 to 0.31], Standard Error of Mean 0.185
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.044, ANCOVA; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.01 to 0.89], Standard Error of Mean 0.214

10. Secondary Outcome: Mean Change From Baseline in Leicester Cough Questionnaire (LCQ) Social Domain Score
Description: The LCQ is a 19-item questionnaire that assesses cough-related Quality-of-Life. It has three domains (physical, psychological and social). The total score range is 3-21 and domain scores each range from 1-7; a higher score indicates a better Quality-of-Life. This outcome measure is the mean change from Baseline to Week 4 in the social domain score.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 39 | 39 | 39 | 39
Points | 0.32 (0.885) | 0.54 (0.950) | -0.03 (1.202) | 0.60 (1.068)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.318, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.19 to 0.58], Standard Error of Mean 0.190
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.030, ANCOVA; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.05 to 0.98], Standard Error of Mean 0.228

11. Secondary Outcome: Mean Change From Baseline in 24-hour Cough Frequency
Description: Cough frequency assessed using an ambulatory cough monitoring device (Leicester Cough Monitor)
Time Frame: Week 4
Population: Fewer participants analyzed than assigned to the groups as some had insufficient recordings.
Measure: Geometric Least Squares Mean (Standard Error); unit: Coughs/hour ratio vs baseline
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 32 | 31 | 32 | 32
Coughs/hour ratio vs baseline | 0.93 (1.114) | 1.00 (1.115) | 0.84 (1.113) | 0.87 (1.112)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.438, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.08, 95% CI 2-sided [0.88 to 1.33], Standard Error of Mean 1.105
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.761, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.04, 95% CI 2-sided [0.82 to 1.31], Standard Error of Mean 1.122

12. Secondary Outcome: Mean Change From Baseline in Awake Cough Frequency
Description: Cough frequency assessed using an ambulatory cough monitoring device (Leicester Cough Monitor)
Time Frame: Week 4
Population: Fewer participants analyzed than assigned to the groups as some had insufficient recordings.
Measure: Geometric Least Squares Mean (Standard Error); unit: Awake coughs/hour ratio vs baseline
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 32 | 31 | 32 | 32
Awake coughs/hour ratio vs baseline | 0.95 (1.119) | 1.03 (1.121) | 0.84 (1.122) | 0.87 (1.121)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.449, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.08, 95% CI 2-sided [0.88 to 1.34], Standard Error of Mean 1.108
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.732, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.04, 95% CI 2-sided [0.82 to 1.32], Standard Error of Mean 1.125

13. Secondary Outcome: Mean Change From Baseline in Night-time Cough Frequency
Description: Cough frequency assessed using an ambulatory cough monitoring device (Leicester Cough Monitor)
Time Frame: Week 4
Population: Fewer participants analyzed than assigned to the groups as some had insufficient recordings.
Measure: Geometric Least Squares Mean (Standard Error); unit: Asleep coughs/hour ratio vs baseline
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 31 | 29 | 29 | 29
Asleep coughs/hour ratio vs baseline | 0.79 (1.180) | 0.90 (1.184) | 0.87 (1.149) | 0.85 (1.145)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.400, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.14, 95% CI 2-sided [0.84 to 1.54], Standard Error of Mean 1.161
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.912, ANCOVA; Ratio of Geometric LS Mean Ratios = 0.98, 95% CI 2-sided [0.69 to 1.40], Standard Error of Mean 1.187

14. Secondary Outcome: Mean Change From Baseline in the Number of Coughing Bouts
Description: Cough frequency assessed using an ambulatory cough monitoring device (Leicester Cough Monitor)
Time Frame: Week 4
Population: Fewer participants analyzed than assigned to the groups as some had insufficient recordings.
Measure: Geometric Least Squares Mean (Standard Error); unit: Bouts/hour ratio vs baseline
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 32 | 31 | 32 | 32
Bouts/hour ratio vs baseline | 0.91 (1.089) | 1.00 (1.090) | 0.82 (1.087) | 0.88 (1.087)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.287, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.09, 95% CI 2-sided [0.93 to 1.29], Standard Error of Mean 1.084
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.420, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.08, 95% CI 2-sided [0.90 to 1.29], Standard Error of Mean 1.092

15. Secondary Outcome: Mean Change From Baseline in the Number of Coughs Per Bout
Description: Cough frequency assessed using an ambulatory cough monitoring device (Leicester Cough Monitor)
Time Frame: Week 4
Population: Fewer participants analyzed than assigned to the groups as some had insufficient recordings.
Measure: Geometric Least Squares Mean (Standard Error); unit: Coughs per bout ratio vs baseline
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
Number analyzed (Participants) | 30 | 30 | 32 | 32
Coughs per bout ratio vs baseline | 0.91 (1.027) | 0.92 (1.027) | 0.98 (1.028) | 0.89 (1.028)
Statistical Analysis 1: Comparison: Placebo (10 mg Cohort) vs Orvepitant 10 mg; Test type: Superiority; p = 0.765, ANCOVA; Ratio of Geometric LS Mean Ratios = 1.01, 95% CI 2-sided [0.96 to 1.05], Standard Error of Mean 1.022
Statistical Analysis 2: Comparison: Placebo (30 mg Cohort) vs Orvepitant 30 mg; Test type: Superiority; p = 0.004, ANCOVA; Ratio of Geometric LS Mean Ratios = 0.90, 95% CI 2-sided [0.85 to 0.97], Standard Error of Mean 1.033

ADVERSE EVENTS:
Time Frame: From enrollment until the final study visit, approximately 13 weeks.
Description: Adverse events that started during the wash-out period were assigned to the treatment received during Treatment Period A. Adverse events that started following first dose in Treatment Period B up to end of follow-up were assigned to the treatment received during Treatment Period B.
Arm/Group | Placebo (10 mg Cohort) | Orvepitant 10 mg | Placebo (30 mg Cohort) | Orvepitant 30 mg
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/40 | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/40 | 1/40 | 3/38 | 1/39
Other Adverse Events (participants affected / at risk) | 18/40 | 30/40 | 17/38 | 20/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (10 mg Cohort) (N=40) | Orvepitant 10 mg (N=40) | Placebo (30 mg Cohort) (N=38) | Orvepitant 30 mg (N=39)
Idiopathic pulmonary fibrosis (exacerbation) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — SAE started during the washout period after receiving orvepitant 10 mg so fatal SAE reported in 'Orv 10 mg' arm. However, the participant died while receiving placebo so death reported in the 'Placebo (10 mg cohort)' arm. Not related to study drug.
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to study drug
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Not related to study drug (for both participants/events)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to study drug
Obstructive pancreatitis (secondary to gallstones) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to study drug
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to study drug
Oxygen saturation decreased (due to no oxygen delivery) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to study drug
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (10 mg Cohort) (N=40) | Orvepitant 10 mg (N=40) | Placebo (30 mg Cohort) (N=38) | Orvepitant 30 mg (N=39)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (3) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Interpretation of the pre-specified efficacy analyses was confounded by a significant treatment by period interaction. This appeared related to a marked placebo response in the first (but not second) treatment period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05185089/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT05185089/SAP_001.pdf